CLINICAL TRIAL: NCT03751462
Title: Prediction of Pseudophakodonesis After Uneventful Cataract Surgery
Brief Title: Prediction of Pseudophakodonesis of Intraocular Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pseudophakodonesis
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract; Pseudoexfoliation; Traumatic cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pseudoexfoliation syndrome (Experimental): Patients with pseudoexfoliation syndrome or traumatic cataract will be examined using the Purkinjemeter device concerning IOL wobble, tilt and decentration
  Interventions: Device: Purkinjemeter

INTERVENTIONS:
Device: Purkinjemeter — The Purkinjemeter will be used for assessment of IOL wobbling, tilt and decentration in patients with pseudoexfoliation syndrome or traumatic cataract

SUMMARY:
Compare visual acuity of patients after cataract surgery with implantation of an IOL clinical outcome measure in eyes with and without pseudoexfoliation syndrome or history of ocular trauma.

DETAILED DESCRIPTION:
Cataract surgery ist the most often performed surgery worldwide and with increasing number of patients undergoing surgery, patients' expectations concerning postoperative optical outcomes are growing. In order to achieve an optimal outcome after cataract surgery an adequate intraocular lens (IOL) centration is essential, especially when premium IOLs like aspheric, toric or multifocal IOls are being implanted. This fact has to be kept in mind especially in patients with pseudoexfoliation syndrome (PXF) or with history of blunt ocular trauma, where decentration and subluxation of the IOL is more likely due to a higher incidence of zonular weakness and zonular dialysis.

Additionally, pseudophacodonesis - dangling of the IOL with eye movement - can occur. Decentration, tilt and dangling of the IOL may decrease visual acuity and contrast sensitivity and induce glare and subjective perception of image flickering. Because of the large amount of pseudophakic patients worldwide, decentered and dislocated IOLs may cause a relatively large public health care burden.

Additionally, IOL implantation in eyes with zonular pathology may be technically challenging. Several devices to improve IOL stability in demanding eyes have been developed and may be used in cases lacking sufficient zonular support, such as different capsular tension rings. Another option would be to use special surgical techniques like scleral fixation of the IOL.

In pseudophakic eyes, IOL tilt and decentration may be measured as an indicator for zonular stability. Several techniques have been used to measure IOL decentration and tilt, such as slitlamp examination, retroillumination photography, Scheimpflug imaging and the analysis of purkinje reflexes. Slitlamp examination is a subjective method that allows approximate decentration measurements, but no quantitative tilt measurements. For this measurement the pupil has to be dilated. Scheimpflug imaging also needs a sufficiently dilated pupil to make the optic edge and the posterior surface of the IOL visible. A recently developed purkinje meter was shown to be highly reproducible to assess IOL tilt and decentration. A new version of this purkinje meter can additionally acquire videos of eye movements. Analysis of these dynamic images can detect dangling or "wobbling" of the lens capsule and the IOL.

Patients within this study will be examined on two occasions. Only one additional visit will be necessary as the first examination will take place on the day of the routine pre-operative visit and all measurements will be non invasive. The results will lead to a better understanding of the long-term outcome after implanting IOLs in eyes with pseudoexfoliation syndrome or a ocular trauma.

ELIGIBILITY:
Inclusion Criteria:

* Cataract with the indication for surgery (decrease in visual acuity, blurred vision or glare ) for both groups (study and control group)
* Age 18 and older
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Written informed consent
* Pseudoexfoliation syndrome or history of blunt ocular trauma - for the study group

Exclusion Criteria:

* Pseudoexfoliation syndrome or history of blunt ocular trauma - for the control group
* History of penetrating ocular trauma
* Relevant other ophthalmic diseases that could affect corneal transparency or the ability for fixation
* Any relevant ophthalmic disease leading to limited visual acuity prognosis after cataract surgery
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
IOL wobble | 12 months
  IOL wobble, tilt and decentration will be assessed in patients with PEX or traumatic cataract using the Purkinjemeter device. The smaller the amount of IOL wobble, tilt and decentration, the better the results.

SECONDARY OUTCOMES:
Best corrected distance visual acuity (BCDVA) | 12 months
  BCDVA will be assessed using a ETDRS chart in 4 meters distance. The more words the patient can read, the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided